CLINICAL TRIAL: NCT00393666
Title: Functional Neuroimaging in Childhood Absence Epilepsy
Brief Title: Why Are Patients With Absence Seizures Absent? A Brain Imaging Study
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Hal Blumenfeld, Principal Investigator, Yale University
Other Study IDs: NIH R01 NS055829; HIC # 18514
Record Dates: First submitted 2006-10-23; First posted 2006-10-30 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Childhood Absence Epilepsy
Keywords: Absence; Epilepsy; Seizure; Brain
MeSH Terms: conditions — Epilepsy, Absence; Epilepsy; Seizures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva samples

SUMMARY:
Our study examines which different brain regions are involved in child absence seizures and how they are related to attention and cognition.

DETAILED DESCRIPTION:
The fundamental mechanisms of altered brain function and impaired attention in childhood absence epilepsy (CAE) are not known. Absence seizures consist of brief 5-10 seconds episodes of unresponsiveness, associated with a 3-4 Hz "spike-wave" discharge on electroencephalogram (EEG). CAE affects 10-15% of children with epilepsy. In addition to the deficit during seizures, many children also suffer from milder attention impairment between absence episodes, which may not be due entirely to medications. Impaired attention during and between absence seizures has a major negative impact on patient quality of life due to deficits in school performance, potential for injuries, and social stigma.

Recent studies suggest that impaired cognition in so-called "generalized" absence seizures may, in fact, depend on dysfunction in specific brain networks. Our central hypothesis is: abnormal function in focal brain regions, such as the anterior cingulate/medial prefrontal cortex and medial thalamus, causes impaired attention both during and between seizures in CAE. If confirmed, this may lead to innovative regional therapies targeted at improving impaired attention in CAE. Specifically, we hope to determine which specific cortical and sub-cortical networks are selectively involved when patients show impaired attention. Using simultaneous EEG and functional magnetic resonance imaging (fMRI), we will determine which brain regions are involved in absence seizures while using a continuous performance task (CPT) to test attention vigilance in the same patients. A few neuropsychology tests will then follow. Patients will be reimbursed $100 as well as all travel and parking expenses.

For more information, please visit www.yalecae.com

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of childhood absence epilepsy or juvenile absence epilepsy
* No other serious health problems or neurological problems
* 6 years or older

Exclusion Criteria:

* No history of myoclonic or tonic-clonic seizures

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Pediatric patients diagnosed with absence epilepsy
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2006-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hal Blumenfeld, MD, PhD, Principal Investigator — Yale University; Michiro Negishi, PhD, Study Director — Diagnostic Radiology; R. Todd Constable, PhD, Study Director — Yale University; Jennifer Guo, MS, Study Director — Yale University
Locations (1):
- Yale University School of Medicine, Neurology Department, New Haven, Connecticut, United States